CLINICAL TRIAL: NCT00490789
Title: A Trial of the Efficacy and Safety of Sirolimus(Rapamycin)Therapy for Renal Angiomyolipmoas in Patients With Tuberous Sclerosis Complex and Sporadic Lymphangioleiomyomatosis
Brief Title: Trial of Efficacy and Safety of Sirolimus in Tuberous Sclerosis and LAM
Acronym: TESSTAL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cardiff University (Other)
Collaborators: University of Nottingham (Other); St Georges Hospital Medical School (Unknown); Royal Sussex County Hospital (Other); The Tuberous Sclerosis Association (Other); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Julian R Sampson, Cardiff University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TESSTAL
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Tuberous Sclerosis; Lymphangioleiomyomatosis
Keywords: tuberous sclerosis; lymphangioleiomyomatosis; sirolimus; angiomyolioma; rapamycin; mTOR
MeSH Terms: conditions — Tuberous Sclerosis; Lymphangioleiomyomatosis | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: sirolimus — daily oral sirolimus with dosage individualised by trough blood levels
  Other Names: rapamune; rapamycin

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the mTOR inhibitor sirolimus as a treatment for renal angiomyolipomas in patients with tyberous sclerosis complex or sporadic lymphangioleiomyomatosis.

DETAILED DESCRIPTION:
Inherited mutations of the TSC1 or TSC2 gene cause tuberous sclerosis while acquired (somatic) mutations of either gene are associated with sporadic lymphangioleiomyomatosis (LAM). Renal angiomyolipomas are a feature of both disorders. TSC1 and TSC2 regulate signalling through the mammalian target of rapamycin (mTOR) pathway. Inhibition of mTOR may result in a decrease in size of TSC 1/2 assciated lesions. We are treating patients with tuberous sclerosis or sporadic LAM with the mTOR inhibitor rapamycin in a non-randomised, open label pilot study of safety and efficacy. Change in size of renal angiomyolipomas is the primary end point

ELIGIBILITY:
Inclusion Criteria:

* If female, documentation of negative pregnancy test prior to enrolment.
* Participants, including males, must use an effective form of contraception, whilst taking sirolimus and for twelve weeks after stopping the drug
* One or more renal angiomyolipomata of at least two centimetres or greater in largest diameter
* Adequate renal function :glomerular filtration rate > 40 ml/min
* Clinically definite diagnosis of tuberous sclerosis (modified Gomez criteria) or sporadic LAM (biopsy-proven or compatible high resolution chest CT scan and respiratory function tests.)
* Signed and dated informed consent

Exclusion Criteria:

* History of non-compliance or inability to give informed consent
* Significant haematological or hepatic abnormality (i.e. transaminase levels > 150 i.u./L serum albumin < 30 g/L, haematocrit< 30%, platelets < 100,000/ mm3, adjusted absolute neutrophil count < 1,500/mm3, total WBC < 3,000/ mm3)
* Greater than 1 g proteinuria daily
* Multiple bilateral AMLs, where individual lesions cannot be distinguished
* Renal haemorrhage within preceding year
* In those who have had a renal haemorrhage, known conservatively managed renal aneurysm(s) greater than 10mm
* Patients who have had embolisation for AML(s) within the preceding 6 months
* Patients who are unable to walk 100 metres on the flat
* Continuous requirement for supplemental oxygen
* Patients who have had or are being considered for organ transplant
* Uncontrolled hyperlipidaemia
* Intercurrent infection at initiation of Sirolimus
* Surgery within last 2 months
* Pregnant or lactating women
* Use of an investigational drug within the last 30 days
* Change in anti epileptic drug medication within the last 3 months
* Likely to need vaccination e.g. for travel during the course of the trial (except for influenza vaccine in patients with LAM)
* Current usage of strong inhibitors of CYP3AE ( such as ketoconazole, voriconazole, itraconazole, tilithromycin or clarithromycin) or strong inducers (such as rifampicin or rifabutin)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2005-10; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
longest diameter of renal angiomyolipomas assessed by MRI scan, toxicity graded by National Cancer Institute's Common Terminology Criteria for Adverse Events v3.0 | assessments at baseline and 2,6,12 and 24 months
toxicity graded by National Cancer Institute's Common Terminology Criteria for Adverse Events | throughout study

SECONDARY OUTCOMES:
respiratory function tests (FEV1, FVC, DLCO), cognitive function (memory, executive skills) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Julian R Sampson, DM, Principal Investigator — Cardiff Univeristy
Locations (3):
- United Kingdom (3):
  - University Hospital of Wales, Cardiff, Wales
  - Royal Sussex County Hospital, Brighton
  - City Hospital, Nottingham

REFERENCES:
- [Derived] Davies DM, de Vries PJ, Johnson SR, McCartney DL, Cox JA, Serra AL, Watson PC, Howe CJ, Doyle T, Pointon K, Cross JJ, Tattersfield AE, Kingswood JC, Sampson JR. Sirolimus therapy for angiomyolipoma in tuberous sclerosis and sporadic lymphangioleiomyomatosis: a phase 2 trial. Clin Cancer Res. 2011 Jun 15;17(12):4071-81. doi: 10.1158/1078-0432.CCR-11-0445. Epub 2011 Apr 27. PMID 21525172